CLINICAL TRIAL: NCT07255222
Title: The Effects of a Multimodal Exercise Program on Physical Performance and Muscle Function in Middle-Aged Patients With Type 2 Diabetes: A Multicenter Randomized Controlled Trial
Brief Title: Effects of a Multimodal Exercise Program on Physical Performance and Muscle Function in Middle-aged Patients With T2DM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: yueh chu wu (Other)
Responsible Party: Sponsor-Investigator, yueh chu wu, Diabetes Educator, Chung Shan Medical University
Organization: Chung Shan Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025-A-35
Record Dates: First submitted 2025-09-25; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This is a multicenter randomized controlled trial with two parallel arms: an intervention group and a control group. Participants will be randomly assigned to either group and assessed at baseline, week 6, and week 12.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A Multimodal Exercise Intervention (Experimental): Participants in this group will participate in a 12-week multimodal exercise program. The program includes supervised training sessions, home-based exercises, and digital support. They will also receive a "Diabetes and Muscle Health Handbook" to guide their training. The goal is to evaluate the effectiveness of this program on muscle function, physical performance, and metabolic control.
  Interventions: Behavioral: A Multimodal Exercise Intervention
- control group (No Intervention): Participants in this group will serve as the control for the study. At the beginning of the study, they will only receive a "Nutrition and Muscle Health Education Sheet". They will not participate in the multimodal exercise program and will continue with their usual health management based on existing medical advice.

INTERVENTIONS:
Behavioral: A Multimodal Exercise Intervention — Participants will receive the same leaflet along with a "Diabetes and Muscle Health Handbook" and will take part in a 12-week multimodal exercise program.
  Arms: A Multimodal Exercise Intervention

SUMMARY:
Background Middle-aged individuals with T2DM, especially in Asian populations, face a heightened risk of sarcopenia. This condition leads to a decline in muscle mass and function, which negatively impacts their quality of life. Effective interventions are therefore urgently needed to slow the progression of the disease and mitigate these risks.

Methods

* Study Design: This is a multicenter randomized controlled trial.
* Participants: The study plans to recruit 66 adults, aged 45 to 64, with a confirmed diagnosis of T2DM.
* Group Assignment: Participants will be randomly assigned to either a control group or an intervention group.

  * Control Group: Participants will receive only a "Nutrition and Muscle Health Education Sheet" and continue with their routine health management based on existing medical advice.
  * Intervention Group: Participants will receive the same leaflet along with a "Diabetes and Muscle Health Handbook" and will take part in a 12-week multimodal exercise program.
* Assessments: All participants will be assessed at baseline, week 6, and week 12.

Outcome Measures

* Primary Outcomes:

  o Physical Function: Short Physical Performance Battery (SPPB), Five-Times Sit-to-Stand Test (5TSTS), handgrip strength, and Skeletal Muscle Mass Index (SMI).
* Secondary Outcomes:

  * Metabolic Control: Glycated hemoglobin (HbA1c).
  * Quality of Life: SF-12 Quality of Life questionnaire.
  * Sarcopenia Risk: Evaluated by the SARC-CalF questionnaire. Expected Outcomes This study aims to provide an evidence-based and feasible multimodal exercise prescription for middle-aged adults with T2DM. The findings are expected to support early intervention strategies for healthy aging and serve as a valuable reference for clinical practice and the development of public health policies.

DETAILED DESCRIPTION:
Primary Outcomes

Physical Function:

Physical performance was assessed using the Short Physical Performance Battery (SPPB), which evaluates lower extremity function through three subtests: balance, gait speed, and chair-stand performance. Each component was scored from 0 to 4, with a total score ranging from 0 to 12, where higher scores indicate better physical performance.

The Five-Times Sit-to-Stand Test (5TSTS) was also used to assess lower limb muscle strength and functional mobility. Participants were instructed to rise from a standard chair (seat height 43-45 cm) to a full standing position and return to sitting five consecutive times as quickly as possible without using their arms. The total time required was recorded in seconds, with longer times indicating poorer performance.

Muscle Strength and Mass:

Handgrip strength was measured using a digital dynamometer (e.g., Jamar or equivalent model) as an indicator of upper limb muscle strength. Participants performed the test in a standing position with the arm fully extended at the side and were instructed to exert maximum force for 3-5 seconds. Two trials were performed for each hand, and the highest value (kg) was used for analysis. Low muscle strength was defined according to the Asian Working Group for Sarcopenia (AWGS 2019) criteria (<28 kg for men and <18 kg for women).

Skeletal Muscle Mass Index (SMI) was determined by bioelectrical impedance analysis (BIA; e.g., InBody 720 or equivalent). Appendicular skeletal muscle mass (ASM, kg) was calculated as the sum of lean mass from both arms and legs. SMI was expressed as ASM divided by height squared (kg/m²). Low muscle mass was defined according to the AWGS 2019 cut-off values (<7.0 kg/m² for men and <5.7 kg/m² for women).

Secondary Outcomes

Metabolic Control:

Glycemic control was evaluated by measuring glycated hemoglobin (HbA1c) levels. Venous blood samples were collected after an overnight fast and analyzed using a standardized high-performance liquid chromatography (HPLC) method. HbA1c values were expressed as percentages according to the National Glycohemoglobin Standardization Program (NGSP) guidelines.

Quality of Life:

Health-related quality of life was assessed using the 12-Item Short Form Health Survey (SF-12). This validated questionnaire consists of 12 items covering eight domains, which are summarized into two composite scores: the Physical Component Summary (PCS) and Mental Component Summary (MCS). Scores were calculated according to the standard scoring manual, with higher scores representing better quality of life.

Sarcopenia Risk Assessment:

Risk of sarcopenia was screened using the SARC-CalF questionnaire, which combines the five-item SARC-F (strength, assistance in walking, rising from a chair, climbing stairs, and falls) with calf circumference measurement. Each item of SARC-F was scored from 0 to 2, yielding a total score ranging from 0 to 10. Calf circumference was measured at the widest point of the right leg using a non-elastic tape, with values ≤34 cm for men and ≤33 cm for women, adding 10 points to the SARC-F score. A total SARC-CalF score ≥11 indicated a high risk of sarcopenia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 2 Diabetes Mellitus and on stable oral hypoglycemic medication.

Middle-aged adults between 45 and 64 years old.

Able to communicate in Mandarin or Taiwanese.

Willing to provide informed consent or have informed consent obtained from a proxy

Exclusion Criteria:

* Limited limb or joint function (e.g., fractures or dislocations).
* Communication or emotional issues, such as depression or mental illness.
* Severe cognitive impairment, such as dementia.
* End-stage renal disease.
* Major comorbidities or complications, including diabetic foot, amputation, myocardial infarction, autonomic neuropathy, and a history of stroke within the last 3 years.

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Short Physical Performance Battery (SPPB) | All participants will be assessed at baseline, week 6, and week 12.
  Physical performance was assessed using the Short Physical Performance Battery (SPPB), which evaluates lower extremity function through three subtests: balance, gait speed, and chair-stand performance. Each component was scored from 0 to 4, with a total score ranging from 0 to 12, where higher scores indicate better physical performance.
Five-Times Sit-to-Stand Test (5TSTS) | All participants will be assessed at baseline, week 6, and week 12.
  The Five-Times Sit-to-Stand Test (5TSTS) was also used to assess lower limb muscle strength and functional mobility. Participants were instructed to rise from a standard chair (seat height 43-45 cm) to a full standing position and return to sitting five consecutive times as quickly as possible without using their arms. The total time required was recorded in seconds, with longer times indicating poorer performance.
Handgrip strength | All participants will be assessed at baseline, week 6, and week 12.
  Handgrip strength was measured using a digital dynamometer (e.g., Jamar or equivalent model) as an indicator of upper limb muscle strength. Participants performed the test in a standing position with the arm fully extended at the side and were instructed to exert maximum force for 3-5 seconds. Two trials were performed for each hand, and the highest value (kg) was used for analysis. Low muscle strength was defined according to the Asian Working Group for Sarcopenia (AWGS 2019) criteria (<28 kg for men and <18 kg for women).
Skeletal Muscle Mass Index (SMI) | All participants will be assessed at baseline, week 6, and week 12.
  Skeletal Muscle Mass Index (SMI) was determined by bioelectrical impedance analysis (BIA; e.g., InBody 720 or equivalent). Appendicular skeletal muscle mass (ASM, kg) was calculated as the sum of lean mass from both arms and legs. SMI was expressed as ASM divided by height squared (kg/m²). Low muscle mass was defined according to the AWGS 2019 cut-off values (<7.0 kg/m² for men and <5.7 kg/m² for women).

SECONDARY OUTCOMES:
Metabolic Control | All participants will be assessed at baseline, week 6, and week 12.
  glycated hemoglobin (HbA1c)

OTHER OUTCOMES:
12-Item Short Form Health Survey (SF-12) | All participants will be assessed at baseline, week 6, and week 12.
  Health-related quality of life was assessed using the 12-Item Short Form Health Survey (SF-12). This validated questionnaire consists of 12 items covering eight domains, which are summarized into two composite scores: the Physical Component Summary (PCS) and Mental Component Summary (MCS). Scores were calculated according to the standard scoring manual, with higher scores representing a better quality of life.
Sarcopenia Risk Assessment | All participants will be assessed at baseline, week 6, and week 12.
  Risk of sarcopenia was screened using the SARC-CalF questionnaire, which combines the five-item SARC-F (strength, assistance in walking, rising from a chair, climbing stairs, and falls) with calf circumference measurement. Each item of SARC-F was scored from 0 to 2, yielding a total score ranging from 0 to 10. Calf circumference was measured at the widest point of the right leg using a non-elastic tape, with values ≤34 cm for men and ≤33 cm for women, adding 10 points to the SARC-F score. A total SARC-CalF score ≥11 indicated a high risk of sarcopenia.

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No